CLINICAL TRIAL: NCT04990115
Title: Bacterial Reduction and Post Operative Pain After Cleaning and Shaping of Root Canals With Single File Systems Used in Different Kinematics
Brief Title: Bacterial Reduction and Post Operative Endodontic-pain Using Different Kinematics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shehab El Din Mohamed Saber, professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-RECD091615
Record Dates: First submitted 2021-06-26; First posted 2021-08-04 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Root Canal Infection
Keywords: Reciprocation; Kinematics; Bacterial reduction; post-operative pain; endodontic flare-ups
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The trial design is a prospective, parallel, randomized with an allocation ratio (1:1), double-blinded, single-center clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Sequentially generated numbers were placed in opaque envelopes until the intervention was conducted and each participant was asked to select an envelope that determine which group of intervention was assumed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotation (Active Comparator): root canal preparation performed using rotating instruments
  Interventions: Other: root canal shaping
- reciprocation (Active Comparator): root canal preparation performed using reciprocating instruments
  Interventions: Other: root canal shaping

INTERVENTIONS:
Other: root canal shaping — root canal treatment

SUMMARY:
This study was conducted to compare the antibacterial effect and degree of postoperative pain of single rotary and reciprocating file systems during endodontic therapy

DETAILED DESCRIPTION:
Introduction: Instrumentation kinematic is one of the many aspects of shaping files that underwent heavy development through the last decade. The impact of the type of motion used to drive shaping instruments was heavily studied but mostly in-vitro. More randomized clinical trials are needed to achieve a reliable body of data concerning the issue.

Aim: This study aimed to evaluate the effect of varying shaping files' kinematics on bacterial reduction, post-operative pain and the incidence of flare-ups. Methods: Necrotic, asymptomatic, single-rooted mandibular premolars with single canals were used in the study, where 46 patients were randomly allocated to two groups. In the first group, WaveOne Gold was used for mechanical preparation while One Shape was used in the second group. Samples were taken preoperatively (S1) and after chemomechanical preparation (S2). Bacterial reduction was evaluated and compared between both groups via culturing technique and quantitative analysis by real-time polymerase chain reaction (qPCR). Post-operative pain and the incidence of flare-ups were also evaluated using the visual analog scale (VAS) method.

ELIGIBILITY:
Inclusion Criteria:

* mandibular premolars
* single rooted
* single canalled
* necrotic pulps
* asymptomatic apical periodontitis

Exclusion Criteria:

* gross caries
* root/crown fracture
* sinus tract
* swelling
* intake of antibiotics within previous 3 months
* pain with percussion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
bacterial reduction | up to 1 hour
  pre-instrumentation and post-instrumentation bacterial cultures to detect change in bacterial count after root canal instrumentation with the different kinematics
post operative pain | after the treatment visit by 24 hours
  Visual analogue scale from 0-100 where 0 is the lowest and 100 is the highest
post operative pain | after the treatment visit by 48 hours
  Visual analogue scale from 0-100 where 0 is the lowest and 100 is the highest
post operative pain | after the treatment visit by 72 hours
  Visual analogue scale from 0-100 where 0 is the lowest and 100 is the highest

CONTACTS AND LOCATIONS:
Overall Officials: shehabeldin M Saber, phd, Principal Investigator — professor
Locations (1):
- Faculty of Dentistry. Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No